CLINICAL TRIAL: NCT03513796
Title: Evaluation of Multiple HCV Diagnosis Pathways for Efficacy, Cost Effectiveness and Cure, in a Regionally Defined General Population
Brief Title: Evaluation of Multiple HCV Diagnosis Pathways for Efficacy, Cost Effectiveness and Cure in NHS Tayside
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016CO01
Record Dates: First submitted 2018-03-27; First posted 2018-05-02 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EVERYONES HCV is a retrospective review of all previous Hepatitis C (HCV) testing and diagnosis in NHS Tayside. The aim of this study is to analyse and compare the different Hepatitis C diagnostic pathways with a view to determining the most cost effective combination of methods of diagnosing HCV infection in a typical developed world population.

DETAILED DESCRIPTION:
Hepatitis C is a blood-borne virus (HCV) that can seriously damage the liver and is spread mainly through blood-to-blood contact with an infected person. The "serious and significant public health risk" posed by HCV was recognised during a member's debate in the Scottish Parliament in 2004. By December 2006, Health Protection Scotland estimated that 50,000 persons in Scotland had been infected with the Hepatitis C virus and that 38,000 were chronic carriers. Currently, the greatest risk of acquiring the virus in the UK is through injecting drug use. In Scotland, it is estimated that over 85% of individuals who have Hepatitis C were infected in this way.

Scotland has taken the lead within the UK in tackling HCV with its Hepatitis C Action Plan. One of the plan's key goals was to identify undiagnosed infections. The plan has identified that access to testing was a significant obstacle in diagnosis. Nearly 75% of undiagnosed cases of HCV within Scotland (16,300) are people who inject drugs (PWIDs) who no longer inject. Given that we have now entered the new era of the curative direct antiviral agents against HCV, it is important that we develop new stratagems to identify and treat those cases

The investigators had considered population screening, however this is not justified under World Health Organisation (WHO) criteria due to the relatively low prevalence in Scotland. The way forward will be to prioritise strategies and target different population groups in a logical manner. The question is what is the most cost-effective means to achieve this and with what combination of testing strategies. Tayside has been at the forefront of piloting novel testing methods. The following list includes the current diagnostic pathways which are standard care in NHS Tayside and previously published pilot studies.

1. Standard diagnosis pathway: clinical suspicion at presentation in primary (pathway 1a) or secondary care (pathway 1b) that HCV could be the cause of the presentation or co-incident issue requiring testing
2. Patients on opiate substitution therapy (OST): testing is being done across the Tayside Substance Misuse Services on initial assessment and annually thereafter.
3. Patients on opiate substitution therapy (OST). Opportunistic testing done for clients receiving OST in participating dispensing pharmacies.
4. Testing in needle exchanges
5. Patients previously on OST or in drug treatment: review of methadone prescription records, dating back to the 1980s, to identify patients at increased risk of HCV
6. Prisons: opt-out testing upon entry is standard practice for all prisoners in the region
7. Community outreach to ethnic minorities, including testing in the mosques
8. General Practice: Electronic record trawl and health promotion

   1. Record trawl with specially designed search tools to identify patients at increased risk of HCV infection and GP follow up offer of testing.
   2. Health promotion message and easy access HCV testing for selected general practices in Tayside.
9. Targeted General Practice screening in Glasgow:

   1. Targeting to GPs in areas with high social deprivation, as these are associated with higher HCV prevalence
   2. Targeting to GPs with in areas with high social deprivation, with patients who have a history of IVDU and fall within the ages of 30-64
10. GP record unification. 24 general practices in Tayside unified their HCV testing records with the secondary care HCV records to identify patients never referred or lost to follow up. Whilst this is not a novel diagnosis pathway, the outcomes will provide important information regarding linkage to care for other pathways.

The investigators intend to retrospectively compare and evaluate the existing and pilot studies that have been conducted in NHS Tayside along with two general practice based studies from Glasgow to determine the optimum and most cost effective bundle of diagnostic activities to bring the different HCV communities to diagnosis and accessing of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All individuals in NHS Tayside tested for Hepatitis C (HCV) between 1st January 1999 and 31st January 2018

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals tested for Hepatitis C (HCV) in NHS Tayside between 1st January 1999 and 31st January 2018
Sampling Method: Probability Sample
Enrollment: 1949 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
Number of HCV tests processed in NHS Tayside between 1999 and 2017 | 16 months
  Total number of HCV IgG and PCR tests processed by NHS Tayside Virology lab between 1999 and 2017

SECONDARY OUTCOMES:
Number of HCV tests that are positive in NHS Tayside between 1999 and 2017 | 16 months
  The number of positive HCV IgG and PCR blood tests processed by NHS Tayside between 1999 and 2017
Number of positive HCV tests by requesting source between 1999 and 2017 | 16 months
  The number of positive HCV tests in NHS Tayside in each requesting healthcare environment.
Cost of HCV testing in each requesting healthcare environment. | 16 months
  The cost of requesting, performing and processing a HCV IgG and PCR test for each healthcare environment.

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, MD, Principal Investigator — University of Dundee and NHS Tayside
Locations (1):
- NHS Tayside, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No